CLINICAL TRIAL: NCT00384449
Title: The Use of a VEGF Inhibitor (Lucentis) in Refractory Macular Edema Due to Eales' Disease
Brief Title: Lucentis (Ranibizumab) for Eales' Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Christina Flaxel, Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF3849s
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Eales' Disease
Keywords: Eales
MeSH Terms: conditions — Eales disease | interventions — Ranibizumab

ARMS (1):
- Lucentis (ranibizumab) (Experimental): Lucentis (ranibizumab)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Consented, enrolled subjects will receive open-label intravitreal injections of 0.5 mg ranibizumab administered once a month for 3 months
  Other Names: Lucentis

SUMMARY:
The primary objective of this protocol is to look at whether Lucentis (ranibizumab) is safe and effective when used for macular edema (retinal swelling) due to Eales' disease. The secondary objective is to see if macular edema comes back within three months after the last dose of study drug is given.

DETAILED DESCRIPTION:
This is a six-month study. Eligible subjects will receive one injection of the study drug into one eye for each of three months. Visual acuity, blood pressure and eye pressure will be tested. Subjects' retinas will be examined and thickness measured by optical coherence tomography (OCT). Safety visits will be scheduled for the week after the injections. The investigators will monitor the subjects' eyes for infection and inflammation. After the three-month treatment period, subjects will return to the clinic monthly for four follow-up visits. Procedures and tests that will be performed at the follow-up visits include visual acuity, a retinal exam including OCT, blood pressure, and eye pressure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study.
* Age > 21 years.
* Disease related considerations:
* For both treatment naïve and previously treated patients:

  * exclusion of all other causes of cystoid macular edema and retinal nonperfusion including branch or central vein occlusion, diabetic retinopathy, sickle retinopathy, sarcoidosis, systemic lupus and other collagen vascular diseases
  * chronic cystoid macular edema as noted clinically and on OCT 3 testing with persistent loss of visual acuity for 3 months or longer
  * if the eye has received prior treatment (including laser photocoagulation and steroids) a 30 day washout period will be required prior to treatment with Lucentis.
* BCVA using ETDRS charts of 20/40 to 20/400 (Snellen equivalent) in the study eye.
* OCT 3 central subfield > or = 250 on 2 separate readings in the central subfield.
* Only one eye will be assessed in the study. If both eyes are eligible, the investigator will determine which eye will be entered into the study.

Exclusion Criteria:

* Treatment for macular edema with intravitreal steroid or macugen within 30 days prior to enrollment in this study.
* Previous vitrectomy within the past 6 months.
* Previous cataract surgery within the preceding 12 months.
* Active intraocular inflammation in the study eye.
* Current vitreous hemorrhage in the study eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Participation in an investigational trial within 30 days of randomization that involved.
* Treatment with any drug that has not received regulatory approval at the time of study entry.
* Known allergy to any component of the study drug.
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
* If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
* Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months. Major surgery is defined as a surgical procedure that is more extensive than fine needle biopsy/aspiration, placement of a central venous access device, removal/biopsy of a skin lesion, or placement of a peripheral venous catheter.
* Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 6 months prior to randomization.
* Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomization.
* Systemic anti-VEGF or pro-VEGF treatment used during the 6 months of the study.
* Current treatment for active systemic infection.
* History of recurrent significant infections or bacterial infections.
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 6 months of the study.
* Subjects meeting any of the following criteria will be excluded from the study:

  * Pregnancy (positive pregnancy test).
  * Prior enrollment in the study.
  * Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
  * Participation in another simultaneous medical investigation or trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina J. Flaxel, MD, Principal Investigator — Casey Eye Institute, Oregon Health & Science University
Locations (1):
- Casey Eye Institute, Portland, Oregon, United States

REFERENCES:
- [Result] Gupta SR, Flaxel CJ. The use of a vascular endothelial growth factor inhibitor (ranibizumab) in macular edema due to eales disease. Retin Cases Brief Rep. 2012 Winter;6(1):122-4. doi: 10.1097/ICB.0b013e31821608e8. PMID 25390730

RESULTS

PARTICIPANT FLOW:
Groups:
- Lucentis (Ranibizumab): Three monthly intravitreal injections of 0.5 mg ranibizumab
Period: Overall Study
Arm/Group | Lucentis (Ranibizumab)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lucentis (Ranibizumab)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in OCT Thickness.
Time Frame: Baseline and 6 months
Population: A patient was enrolled, but then became ineligible. The same patient was later re-enrolled and maintained eligibility.
Measure: Number; unit: um
Arm/Group | Lucentis (Ranibizumab)
Number analyzed (Participants) | 1
um
  Baseline, Day 0 | 269
  Month 6 | 262

2. Primary Outcome: Incidence and Severity of Ocular Adverse Events, as Identified by Eye Examination (Including Visual Acuity Testing)
Time Frame: Monthly through Month 6
Population: A patient was enrolled, but then became ineligible. The same patient was later re-enrolled and maintained eligibility.
Measure: Number; unit: adverse events
Arm/Group | Lucentis (Ranibizumab)
Number analyzed (Participants) | 1
adverse events | 0

3. Primary Outcome: Incidence and Severity of Other Adverse Events, as Identified by Physical Examination, Subject Reporting, and Changes in Vital Signs
Description: No adverse events.
Time Frame: Monthly through Month 6
Population: A patient was enrolled, but then became ineligible. The same patient was later re-enrolled and maintained eligibility.
Measure: Number; unit: adverse events
Arm/Group | Lucentis (Ranibizumab)
Number analyzed (Participants) | 1
adverse events | 0

4. Secondary Outcome: BCVA, as Assessed by the Number of Letters Read Correctly on the ETDRS Eye Chart at a Starting Test Distance of 4 Meters.
Time Frame: Months 3,4,5 and 6
Population: A patient was enrolled, but then became ineligible. The same patient was later re-enrolled and maintained eligibility.
Measure: Number; unit: letters
Arm/Group | Lucentis (Ranibizumab)
Number analyzed (Participants) | 1
letters
  Month 3 | 63
  Month 4 | 70
  Month 5 | 64
  Month 6 | 60

5. Secondary Outcome: Incidence of Ocular and Non-ocular Adverse Events Evaluated Through Month 6.
Description: No adverse events.
Time Frame: Monthly through Month 6
Measure: Number; unit: adverse events
Arm/Group | Lucentis (Ranibizumab)
Number analyzed (Participants) | 1
adverse events | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Lucentis (Ranibizumab): Three monthly intravitreal injections of 0.5 mg of ranibizumab
Arm/Group | Lucentis (Ranibizumab)
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes